CLINICAL TRIAL: NCT00990093
Title: A Randomised, Cross-over, Open-labelled Study Evaluating the Acceptance of Test Catheters Compared to SpeediCath Catheters
Brief Title: A Randomised, Cross-over, Open-labelled Test Catheter Acceptance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP062CC
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Intermittent Urethral Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- test intermittent catheter (Experimental): CH 12 hydrophilic coated catheter
  Interventions: Device: test intermittent catheter
- intermittent catheter (Experimental): CH 12 hydrophilic coated catheter
  Interventions: Device: Intermittent catheterization

INTERVENTIONS:
Device: test intermittent catheter — CH 12 hydrophilic coated catheter
  Other Names: Test catheter
  Arms: test intermittent catheter
Device: Intermittent catheterization — CH 12 hydrophilic catheter
  Other Names: SpeediCath
  Arms: intermittent catheter

SUMMARY:
The purpose of this study is to evaluate that the test catheter is no less accepted than the SpeediCath (SC) catheter.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Has normal/impaired sensation in the urethra
* Self-catheterises at least 4 times per day
* Has used clean self-intermittent catheterisation for at least 14 days
* Is able to open and prepare the catheters for catheterisation
* Has signed the informed consent before any study related-activities.

Exclusion Criteria:

* Has a symptomatic urinary tract infection as assessed by the investigator
* Is mentally unstable as assessed by the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fin Biering-Sørensen, MD, Principal Investigator — Klinik for Rygmarvsskader, Rigshospitalet
Locations (1):
- Klinik for Rygmarvsskader, Hornbæk, Denmark

REFERENCES:
- [Derived] Prieto JA, Murphy CL, Stewart F, Fader M. Intermittent catheter techniques, strategies and designs for managing long-term bladder conditions. Cochrane Database Syst Rev. 2021 Oct 26;10(10):CD006008. doi: 10.1002/14651858.CD006008.pub5. PMID 34699062
- [Derived] Chartier-Kastler E, Lauge I, Ruffion A, Goossens D, Charvier K, Biering-Sorensen F. Safety of a new compact catheter for men with neurogenic bladder dysfunction: a randomised, crossover and open-labelled study. Spinal Cord. 2011 Jul;49(7):844-50. doi: 10.1038/sc.2011.5. Epub 2011 Feb 22. PMID 21339763

RESULTS

PARTICIPANT FLOW:
Groups:
- A: First Test Catheter Then Standard Catheter; B: First Standard Catheter Then Test Catheter: Test catheter is a CH 12 hydrophilic coated intermittent catheter
Period: Test Period 1 (1-14 Days)
Arm/Group | A: First Test Catheter Then Standard Catheter | B: First Standard Catheter Then Test Catheter
Started | 19 | 17
Completed | 15 | 15
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 1 | 0
Not completed — Lack of Efficacy | 0 | 2
Period: Test Period 2 (15-28 Days)
Arm/Group | A: First Test Catheter Then Standard Catheter | B: First Standard Catheter Then Test Catheter
Started | 15 | 15
Completed | 13 | 14
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 4
Age Continuous [Median (Full Range); unit: years] | 43.2 [20.0 to 69.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Region of Enrollment [Number; unit: participants]
  Denmark | 24
  France | 12

OUTCOME MEASURES:

1. Primary Outcome: Discomfort Measured on a VAS Scale 0 Being no Discomfort, 10 Being Worst Imaginable Discomfort.
Description: Participants were to test the catheter by self-catheterising a minimum of 4 catheters each day for 14 days.
  At the end of each study period participants were asked to indicate how they would rate the discomfort experienced during the catheterisation procedures. Discomfort was measured by the participants own rating of discomfort on a VAS scale from 0 (no discomfort) to 10 (worst imaginable discomfort)
Time Frame: 14 days
Population: Six participants discontinued the study in the first test period, i.e. before visit 2 at which the first catheter evaluation was to be given. The primary outcome was the catheter evaluation on discomfort, and these six participants did not contribute to the ITT analysis of the primary outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test Catheter: SpeediCath Compact Male Catheter
- Standard Catheter: SpeediCath Catheter
Arm/Group | Test Catheter | Standard Catheter
Number analyzed (Participants) | 30 | 30
units on a scale | 1.59 (2.28) | 1.94 (2.24)

ADVERSE EVENTS:
Groups:
- Test Catheter: SpeediCath Compact Male
- Standard Catheter: SpeediCath, CH 12 hydrophilic coated intermittent catheter
Arm/Group | Test Catheter | Standard Catheter
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 1/32 | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Catheter (N=32) | Standard Catheter (N=34)
epididymitis (Infections and infestations) | 0 | 1
discomfort during insertion (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less